CLINICAL TRIAL: NCT05707520
Title: Clinical Evaluation of the Long-term Benefit of Enteric-coated Mycophenolate (MPAs) After Liver Transplantation
Brief Title: Long-term Benefit of MPA in Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other); RenJi Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Beijing YouAn Hospital (Other); Huashan Hospital (Other); The Third Xiangya Hospital of Central South University (Other); West China Hospital (Other); Hebei Medical University Third Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Beijing Friendship Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yang Yang, Vice president of third Affiliated Hospital, Sun Yat-Sen University, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2022]02-146-01
Record Dates: First submitted 2023-01-06; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Liver Transplant Rejection; Immunosuppressant Adverse Reaction
Keywords: enteric-coated mycophenolate; adverse reaction; liver transplantation; transplant rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPA: Immunosuppressant with enteric-coated mycophenolate sodium
  Interventions: Drug: enteric-coated mycophenolate (MPAs)
- None MPA: Immunosuppressant without enteric-coated mycophenolate sodium
  Interventions: Drug: None MPA

INTERVENTIONS:
Drug: enteric-coated mycophenolate (MPAs) — Immunosuppression protocol with enteric-coated mycophenolate sodium
  Groups: MPA
Drug: None MPA — Immunosuppression protocol without enteric-coated mycophenolate sodium
  Groups: None MPA

SUMMARY:
MPA drugs are antiproliferative immunosuppressants and are widely used in solid organ transplantation. MPA drugs do not affect the recipient's kidney function and do not cause metabolic abnormalities and other problems. Intestinal solvent-based MPA drugs are widely used in clinical practice by improving the dosage form, reducing the irritation of MPA to the mucosa of the digestive tract, improving the tolerability of patients and maintaining a sufficient amount of MPA. However, data on the use/long-term use of intestinal solvent-based MPAs in liver transplant recipients are lacking. The study aims to evaluate the long-term benefits of enteric-coated mycophenolic acid in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent their first liver transplantation between January 1, 2016 and February 28, 2021;
* Recipient's survival time≥ 1 year;
* Age 18~65 years old;
* Patients with complete data and no loss to follow-up.

Exclusion Criteria:

* use of other types of anti-metabolic immunosuppressants;
* Second liver transplantation for various reasons within 1 year after the first transplantation;
* Patients with serious underlying diseases, including heart disease, infection and renal insufficiency, combined with other malignant tumors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long-term survived liver transplant recipients in 13 hospitals in China
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
complex endpoint | 60 months after liver transplantation
  Graft loss or reoccurrence of HCC, or neoplasm, or death

SECONDARY OUTCOMES:
Late onset acute rejection | 60 months after liver transplantation
  rejection diagnosed by liver test, pathologic diagnosis by biopsy
Incidence of AKI or CKD | 60 months after liver transplantation
  AKI/CKD diagnosed according to KDIGO 2012 AKI and CKD diagnosis criteria
Adverse events | 60 months after liver transplantation
  Incidence of leukopenia/neutropenia, incidence of viral infections, incidence of new tumors (non-liver cancer).

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data will be shared on ResMan, after completion and the consent from investigators and IRB